CLINICAL TRIAL: NCT06810778
Title: Phase I/II Study of Duvelisib and Venetoclax in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Brief Title: Duvelisib and Venetoclax in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma (PTCL)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-001373; NCI-2025-00574 (Registry Identifier: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2025-01-24; First posted 2025-02-06 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: T-cell-prolymphocytic Leukemia; Cutaneous T-Cell Lymphoma Refractory
Keywords: leukemia; refractory; relapsed
MeSH Terms: conditions — Leukemia, Prolymphocytic, T-Cell; Leukemia; Recurrence | interventions — duvelisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm Treatment (Duvelisib and Venetoclax) (Experimental): Phase I:
  In the phase I study, 2 dose levels of duvelisib (15 and 25 mg BID) and 3 dose levels of venetoclax (200, 400, and 800 mg QD) will be evaluated. Patients will start with 15 mg BID of duvelisib and 200 mg QD of venetoclax. We use a traditional 3 + 3 design to accrue patients to each combination cohort. There are 5 possible dosing combinations to be tested, with up to 18 patients planned to be enrolled. Enrollment may stop early based on DLTs. The DLT assessment window is defined as Day 1-21 of Cycle 1 (21 days). De-escalation will occur if unexpected toxicity is observed and both drugs will be reduced for the next lower dosing cohort. Increasing drug dosing levels will be performed in parallel cohorts, each increasing either venetoclax or duvelisib.
  Interventions: Drug: Duvelisib; Drug: Venetoclax

INTERVENTIONS:
Drug: Duvelisib — 15 and 25 mg BID
Drug: Venetoclax — 200, 400, and 800 mg QD

SUMMARY:
This is an open-label, phase I/II study of duvelisib in combination with Venetoclax for patients with relapsed/refractory NHL. Duvelisib is an FDA approved, marketed product used to treat certain patients with leukemia and lymphoma and Venetoclax, which is approved for treatment of certain patients with acute myeloid leukemia. The combination of these two drugs is experimental. Experimental means that it is not approved by the United States Food and Drug Administration (FDA). The researchers want to find out how safe it is to combine these drugs and how well this combination can work for your cancer.

DETAILED DESCRIPTION:
In this phase I/II trial, we combine duvelisib and venetoclax in patients with relapsed/refractory Peripheral T-cell lymphoma (PTCL). Researchers aim to determine the maximum tolerated doses (MTD) of duvelisib in combination with venetoclax, the safety of combination therapy, and preliminary efficacy data in Peripheral T-cell lymphoma (PTCL).

Patients with PTCL would be offered the option to remain on treatment beyond 2 years if they are clinically benefitting, complete response, partial response, stable disease (CR, PR, SD).

The phase I portion of the trial will determine the dose, schedule, safety, and tolerability of duvelisib in combination with venetoclax.

Phase I:

In the phase I study, 2 dose levels of duvelisib (15 and 25 mg BID) and 3 dose levels of venetoclax (200, 400, and 800 mg QD) will be evaluated. Patients will start with 15 mg BID of duvelisib and 200 mg QD of venetoclax. We use a traditional 3 + 3 design to accrue patients to each combination cohort. There are 5 possible dosing combinations to be tested, with up to 18 patients planned to be enrolled. Enrollment may stop early based on DLTs. The DLT assessment window is defined as Day 1-21 of Cycle 1 (21 days). De-escalation will occur if unexpected toxicity is observed and both drugs will be reduced for the next lower dosing cohort. Increasing drug dosing levels will be performed in parallel cohorts, each increasing either venetoclax or duvelisib (see Dosing Schema).

The following lymphoma subtypes will be excluded due to potential tumor lysis risk: cutaneous T-cell lymphoma (CTCL) and T-cell-prolymphocytic leukemia (TPLL).

Patients in the initial dosing cohorts will start at a lower dose of venetoclax than the tested dose in phase 2 trials dose (800 mg QD) and at a lower dose of duvelisib than the recommended phase 2 dose (25 mg BID). Once the RP2D of combination duvelisib plus venetoclax is determined, patients assigned to lower dose levels in the phase I trial will have the option to escalate their duvelisib and venetoclax doses to the RP2D.

Planned Phase II (dependent on phase I data and new discussions with AbbVie and Secura Bio):

The phase II study will only proceed after discussion of Phase I results with study investigators, DSMB, AbbVie, and Secura Bio and will enroll patients with relapsed/refractory PTCL at the RP2D.

Phase II will start once phase I data have been reviewed by AbbVie and Secura Bio, DSMB, and FDA, and proceeding to the next phase has been approved.

Study visits will occur weekly through cycles 1-2, once per cycle during cycles 3-7, every 2 cycles from cycle 8-13, and every 3 cycles thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Histologically confirmed relapsed/refractory PTCL, except the following lymphoma subtypes: cutaneous T-cell lymphoma (CTCL) and T-cell-prolymphocytic leukemia (TPLL).
* Phase II: same as phase I
* Disease that has progressed during or relapsed after at least two previous therapies.
* ECOG performance status ≤ 2
* Adequate hepatic function defined as:

  o Serum aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x upper limit of normal (ULN), bilirubin ≤ 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin
* Adequate renal function as defined by:

  o Creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection
* Patients must meet the following hematologic criteria at screening, unless they have significant bone marrow involvement confirmed on biopsy:

  * Absolute neutrophil count ≥ 1500 cells/mm3 (1.5 x 109/L) or ≥ 1000 cells/mm3 (1.5 x 109/L) with bone marrow involvement. Growth factor use is allowed in order to achieve this
  * Platelet count ≥ 50,000 cells/mm3 (50 x 109/L) independent of transfusion within 7 days of screening
  * Hemoglobin ≥8 g/dL (without transfusion support.)

Exclusion Criteria:

* Phase I and Phase II:

  * Patients eligible for Hematopoietic stem cell transplantation (HSCT)
  * Cutaneous T-cell lymphoma (CTCL) and T-cell-prolymphocytic leukemia (TPLL)
  * Suspected and confirmed central nervous system involvement
  * Previous treatment with venetoclax or a PI3K inhibitor.
  * Active malignancy other than NHL requiring ongoing therapy, with the exception of hormonal therapy (i.e. castration-sensitive prostate cancer stable on testosterone blockade)
  * Patients receiving cancer therapy (i.e., chemotherapy, radiation therapy, immunotherapy, biologic therapy, surgery) within 2 weeks of Cycle 1/Day 1 with the following exceptions:

    * For patients on targeted therapies, a washout of least five half-lives is required
    * Patients who experience clinical deterioration may start therapy after a shorter washout period with prior approval by the PI
    * Corticosteroid therapy (prednisone or equivalent <20 mg daily) is allowed
    * Patients with multiple basal cell carcinomas that undergo sequential Moh's excisions with interim observation
  * Allogeneic hematologic stem cell transplant within 6 months of starting study treatment or active graft vs. host disease (GVHD) requiring treatment or prophylaxis

    o Patients with a history of an allogeneic stem cell transplant > 6 months prior to starting study treatment should be stable, off of immunosuppression for at least 2 months.
  * Any active systemic infection requiring systemic antibiotics or other uncontrolled, active infections
  * Positive Human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) antibody test

    o For HCV and HBV, patients with evidence of prior infection also excluded
  * Evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    * Uncontrolled and/or active systemic infection (viral, bacterial or fungal)
    * Chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface (HBs) antigen negative-, anti-HBs antibody positive and anti-hepatitis B core (HBc) antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate
  * Uncontrolled, not disease-related autoimmune hemolytic anemia or ITP
  * History of stroke or intracranial hemorrhage
  * History of severe bleeding disorder (hemophilia A or B, von Willebrand disease (VWD)), history of spontaneous bleeding requiring blood transfusions or other medical intervention, history of life-threatening hemorrhage within 3 months of first dose.
  * Currently active gastrointestinal disease, including colitis, inflammatory bowel disease and diarrhea requiring therapy
  * Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to enrollment
  * Cardiac history of CHF requiring treatment or Ejection Fraction ≤ 50% or chronic stable angina
  * Use of Coumadin for anticoagulation (other anticoagulants permitted)
  * Lactating or pregnant
  * Unable to swallow capsules or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction resulting in malabsorption or chronic diarrhea
  * Concurrent administration of medications or foods that are strong inhibitors or inducers of CYP3A (see Appendix D)
  * Treatment with any of the following within 7 days prior to the first dose of study drug:
  * Steroid therapy for anti-neoplastic intent (defined as prednisone or equivalent >20 mg daily)
  * Moderate or strong cytochrome P450 3A (CYP3A) inhibitors (see Appendix D for examples)
  * Moderate or strong CYP3A inducers (see Appendix D for examples)
  * Administration or consumption of any of the following within 7 days prior to the first dose of study drug:

    * Grapefruit or grapefruit products
    * Seville oranges (including marmalade containing Seville oranges)
    * Star fruit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the dose limiting toxicities (DLTs), for the combination regimen of duvelisib plus venetoclax for patients with relapsed or refractory PTCL | Up to 21 days
  Phase I:
  Will be graded according to the Common Terminology Criteria for Adverse Events version 5.0.
Determine the Maximum Tolerated Dose MTD) | Up to 21 days
  Phase I:
  Will be defined as the highest dose studied for which the observed incidence of DLT is less than 33%. Frequencies of toxicities will be tabulated according to the National Cancer Institute Common Toxicity Criteria.
Recommended phase II dose (Phase I) | Up to 21 days
  Phase I

SECONDARY OUTCOMES:
Overall response rate | up to 1 year
  Phase II:
  Will be assessed according to Lugano criteria. Will be based on exact one-sided binomial tests (Simon two-stage designs) within each of the disease groups. Will be estimated with exact 95% confidence intervals.
Objective response rate | Up to 1 year
  Phase II:
  Will be defined as proportion of patients who achieve a complete and partial response. Will be estimated along with a 95% confidence interval
Duration of response | From the date of response to the date of progression of disease, assessed up to 1 year
  Phase II:
  Will be calculated using Kaplan-Meier methodology.
Progression free survival | From start of treatment to the date of progression, death or last follow-up, assessed up to 1 year
  Phase II:
  Will be calculated using Kaplan-Meier methodology.
Overall survival | From the start of treatment to the date of death or last follow-up, assessed up to 1 year
  Phase II:
  Will be calculated using Kaplan-Meier methodology.
Pharmacokinetic parameters: Half-life | At days 1, 8, and 15 of cycle 1 (1 cycle = 21 days)
  Phase II:
  Will include half-life determined using non-compartmental methods. Standard descriptive statistics (mean, standard deviation, median, range) will be presented on all parameters.
Pharmacokinetic parameters: Maximum concentration | At days 1, 8, and 15 of cycle 1 (1 cycle = 21 days)
  Phase II:
  Will include maximum concentration determined using non-compartmental methods. Standard descriptive statistics (mean, standard deviation, median, range) will be presented on all parameters.
Pharmacokinetic parameters: Area under the curve | At days 1, 8, and 15 of cycle 1 (1 cycle = 21 days)
  Phase II:
  Will include area under the curve determined using non-compartmental methods. Standard descriptive statistics (mean, standard deviation, median, range) will be presented on all parameters.
Pharmacokinetic parameters: Volume of distribution | At days 1, 8, and 15 of cycle 1 (1 cycle = 21 days)
  Phase II:
  Will include volume of distribution determined using non-compartmental methods. Standard descriptive statistics (mean, standard deviation, median, range) will be presented on all parameters.
Pharmacokinetic parameters: Clearance | At days 1, 8, and 15 of cycle 1 (1 cycle = 21 days)
  Phase II:
  Will include clearance determined using non-compartmental methods. Standard descriptive statistics (mean, standard deviation, median, range) will be presented on all parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- David Geffen School of Medicine at the University of California at Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided